CLINICAL TRIAL: NCT02472990
Title: Determining Biomechanical and Morphological Factors That Affect Children With Duchenne Muscular Dystrophy (DMD) Who Loss of the Ability to Walk
Brief Title: Biomechanical and Morphological Changes in Dystrophic Muscle
Acronym: MARCHE-DMD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MARCHE-DMD
Record Dates: First submitted 2015-06-10; First posted 2015-06-16 (Estimated); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Duchenne Dystrophy Muscular
Keywords: DMD; morphological predictive factors; Mechanical
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Duchenne muscular dystrophy children (Other): No drug and no placebo were used in this study. For 2h30 (time)
  * Measurement of leg strength using a dynamometer
  * Measurement of Motor Function
  * Walk test 6 minutes
  * Walk test 10 meters
  * Walk analysis: 3D recording of walking
  * Muscle MRI
  Interventions: Other: No drug and no placebo were used in this study
- Healthy children (Other): No drug and no placebo were used in this study. For 2h30 (time)
  * Measurement of leg strength using a dynamometer
  * Measurement of Motor Function
  * Walk test 6 minutes
  * Walk test 10 meters
  * Walk analysis: 3D recording of walking
  * Muscle MRI
  Interventions: Other: No drug and no placebo were used in this study

INTERVENTIONS:
Other: No drug and no placebo were used in this study — measures of muscular strength of legs, motor function, walk testing and analysis (3D video recording), RMI
  Other Names: Several parameters must be performed.

SUMMARY:
The loss of ability to walk in many children with DMD (Duchenne muscular Dystrophy) is a pejorative event. Biomechanical and morphological unknowledge about the loss of the walk ability in children with DMD is an obstacle in reeducative, pharmacological or surgical therapeutic targets.

DETAILED DESCRIPTION:
The loss of ability to walk in many children with DMD (Duchenne muscular Dystrophy) is a pejorative event. Biomechanical and morphological unknowledge about the loss of the walk ability in children with DMD is an obstacle in reeducative, pharmacological or surgical therapeutic targets. We suppose that there are muscular characteristics and predictive parameters of the loss of walk ability. The identification of these potential therapeutic targets would improve the surveillance and the clinical care but would also guide future clinical and fundamental trials too.

ELIGIBILITY:
Inclusion Criteria:

* Young man ou woman (5 to 17 years old) with Duchenne Muscular Dystrophy (confirmed by immunohistochimy on the muscular biopsy and/or mutation in the dystrophin confirmed by molecular biology)
* Time more than 7 secondes to test of 10 m and/or distance less than 330 m to walk test of 6 minutes. These values are recent markers to include children with a strong risk of loss of walking ability in 2 years.
* Parental inform sign consent and / or child inform consent

Exclusion Criteria:

* Recent orthopaedic surgery of lower limbs (6 months)
* Other chronic disease associated, which have an impact on the walking
* Cognitive Deficiency or behavior disorders limiting the understanding of the study
* Children who can benefit ATU (translarna ® or other) during the study
* All MRI contradications : pacemaker or neurosensory stimulator or implantable defibrillator, neurosurgical valves, cochlear implant or ferromagnetic implants near nervous structures, brace, metallic prostheses, not cooperative or agitated patients, patient claustrophobic, pregnant woman.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Determine biomechanical and morphological predictive factors of the loss of the walk ability of the children with DMD | 24 years
  Determine the biomechanical factors (muscular atrophy, muscular strength, muscular shrinkage) and morphological (greasy infiltration, contractile portion, muscular geometry) predictive of the loss of the walk ability of the children with DMD

SECONDARY OUTCOMES:
Identify the muscles wasting and their implication in the loss of strength and the walking ability | 24 years
  Identify the muscles wasting and their implication in the loss of strength and walking. This will be made possible thanks to the predictive analysis and the evolutionary analysis of the MRI and strength before and after loss of walking ability
Biomechanical evolutionary data collected during the last 2 years of walking | 24 years
  Biomechanical evolutionary data collected during the last 2 years of walking by the repetition of the analysis of the walking until the loss of the walking ability.
Establish the relationship between the parameters of walking and the scrawny body morphological anomalies | 24 years
  Establish the relationship between the parameters of walking and the scrawny body morphological anomalies (muscular Atrophy, greasy infiltration, contractile muscular portion, three-dimensional morphological parameters) by doing correlations analysis

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHRU, Brest, Brittanny
  - CHRU, Lille, North
  - CHRU, Angers
  - CH Le Mans, Le Mans
  - CHU, Lyon
  - CHU de Nantes, Nantes
  - CHU, Poitiers
  - CHU, Rennes
  - CHRU, Tours
  - CHBA, Vannes